CLINICAL TRIAL: NCT02578641
Title: A Multicentre, Randomized, Open-Label, Phase III Clinical Trial Of Gemcitabine And Carboplatin Followed By Epstein-Barr Virus-Specific Autologous Cytotoxic T Lymphocytes Versus Gemcitabine And Carboplatin As First Line Treatment For Advanced Nasopharyngeal Carcinoma(NPC) Patients
Brief Title: A Phase III Trial Evaluating Chemotherapy and Immunotherapy for Advanced Nasopharyngeal Carcinoma (NPC) Patients
Acronym: VANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tessa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF01
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma (NPC); NPC; immunotherapy; Nasopharyngeal Cancer; Nose Cancer; Cell therapy; Head and Neck Cancer; Cytotoxic T cells; chemotherapy; Epstein-Barr Virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nose Neoplasms; Head and Neck Neoplasms; Epstein-Barr Virus Infections | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): 4 cycles* of combination IV Gemcitabine (1000 mg/m2) and IV carboplatin (AUC2) on Days 1, 8, 15 every 28 days, followed sequentially by T-cell immunotherapy (2 cycles) of autologous EBV specific Cytotoxic T cells every 2 weeks, followed by EBV-specific CTL immunotherapy (4 cycles) every 8 weeks after 6 weeks from the second cycle.
  *Additional 1-2 chemotherapy cycles (up to total 6 chemo cycles) might be given upon discretion of Investigator, if EBV-specific CTL infusions are not available in time for the 1st scheduled infusion.
  As of 1 May 2020, patients who have not received the first infusion of EBV-specific CTLs, will instead continue to receive a total of 6 cycles combination of Gemcitabine (1000 mg/m2) and carboplatin (AUC2) on Days 1, 8, 15 every 28 days
  Interventions: Biological: autologous EBV specific Cytotoxic T cells; Drug: combination IV gemcitabine and IV carboplatin (AUC2)
- Arm B (Active Comparator): 6 cycles of combination IV gemcitabine (1000 mg/m2) and IV carboplatin (AUC2) on Days 1, 8, 15 every 28 days.
  Interventions: Drug: combination IV gemcitabine and IV carboplatin (AUC2)

INTERVENTIONS:
Biological: autologous EBV specific Cytotoxic T cells — The CTL line will be prepared by co-cultivation of the irradiated EBV-LCL with patient PBMC. A proportion of peripheral blood will be used to generate EBV specific CTLs.
  Arms: Arm A
Drug: combination IV gemcitabine and IV carboplatin (AUC2) — 4 cycles for Arm A and 6 cycles for Arm B

SUMMARY:
This study is a multi-center, randomized, open label, Phase III clinical trial for advanced Nasopharyngeal Carcinoma(NPC) Patients.

Drugs used in chemotherapy, such as gemcitabine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving an infusion of a person's cytotoxic T cells (CTL) that have been treated in the laboratory may help the body build an effective immune response to kill tumor cells. Giving combination chemotherapy together with laboratory-treated T cells may kill more tumor cells. This Phase III trial is to assess if combined gemcitabine-carboplatin (GC) followed by adoptive T-cell therapy would improve clinical outcome for patients with advanced nasopharyngeal carcinoma (NPC). It is also the world's first, and largest, Phase 3 T-cell therapy cancer trial ever conducted, and enrollment is ongoing for 330 patients from 30 hospital centers across Asia and the United States.

This clinical trial is conducted on the back of a successful Phase 2 NPC trial involving 38 patients at the National Cancer Centre, Singapore. This trial produced the best published 2-year (62.9%), and median overall survival (OS) data (29.9 months) in 35 patients with advanced NPC who received autologous EBV-specific CTL. Kindly see https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3978790/ for the Phase 2 publication titled "Adoptive T-cell Transfer and Chemotherapy in the First line treatment of Metastatic and/or Locally Recurrent Nasopharyngeal Carcinoma".

DETAILED DESCRIPTION:
330 patients will be randomized after their eligibility status has been fully determined and informed consent has been obtained. Patients will be randomly allocated to receive either Arm A (Gemcitabine and Carboplatin (GC) x 4* cycles and EBV-specific CTL) or Arm B (GC x 6 cycles alone) in a 1:1 ratio using a stratified block randomization scheme. The stratification variables are country and disease stage (metastatic vs locally recurrent). *Additional 1-2 chemotherapy cycles (up to total 6 chemo cycles) might be given upon discretion of Investigator, if EBV-specific CTL infusions are not available in time for the 1st scheduled infusion.

After randomization, patients in Arm A will have their peripheral blood taken for the establishment of cytotoxic T cell line and EBV transformed lymphoblastoid cell line (CTL). Within two weeks of enrollment, patients will commence combination GC chemotherapy for a total of 4 cycles. Patients in Stage 2 of study will receive the EBV-specific CTL immunotherapy.

As of 1 May 2020, patients who have not received the first infusion of EBV-specific CTLs, will instead continue to receive a total of 6 cycles combination of Gemcitabine (1000 mg/m2) and carboplatin (AUC2) on Days 1, 8, 15 every 28 days

ELIGIBILITY:
Key Inclusion Criteria

1. Metastatic or locally recurrent EBV-positive, non-keratinizing and/ or undifferentiated NPC* who do not have curative options such as chemo-radiation or surgery

   *Subjects will be enrolled based on confirmed histology diagnosis of the NPC
2. Radiologically measurable disease as per RECIST 1.1
3. Human Immunodeficiency Virus (HIV) negative*

   * Status of HIV must be confirmed via a HIV antibody test or other confirmatory tests available within 4 weeks of screening
4. Bilirubin <2 x upper limit of normal (ULN) and aspartate aminotransferase (AST), alanine aminotransferase (ALT) <3 x ULN
5. Calculated creatinine clearance (CRCL) ≥40 mL/min. Glomerular Filtration Rate (GFR) is calculated based on Cockcroft-Gault method.
6. Normal corrected calcium levels
7. Absolute neutrophil count >1200/mm3, hemoglobin (Hb) ≥10 g/dL and platelets ≥100,000/mm3
8. Male or female
9. Age ≥ 18 years or according to local legal age of consent
10. Eastern Cooperative Oncology Group Performance Scale (ECOG-PS) ≤2
11. Written informed consent
12. Life expectancy >6 months

Key Exclusion Criteria

1. Severe concomitant illness i.e. chronic obstructive pulmonary disease (COPD), ischemic heart disease (IHD), active congestive cardiac failure (CCF), active angina pectoris, uncontrolled arrhythmia, uncontrolled hypertension
2. HIV Positive*

   * Status of HIV must be confirmed via a HIV antibody test or other confirmatory tests available within 4 weeks of screening
3. Pregnant or lactating females
4. Refuse of use of contraception during trial (both male and female patients)
5. Investigational therapy less than one month prior to study entry
6. Pre-existing peripheral neuropathy (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] ≥2)
7. Central nervous system metastasis
8. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis and T1] or any cancer curatively treated >3 years prior to study entry
9. Positive hepatitis B surface antigen (HBsAg) results
10. Known history of hepatitis C and recovery status has not been determined at time of screening
11. Prior anti-cancer treatment for metastatic or locally recurrent disease, EXCEPT:

    For metastatic or locally recurrent disease, localised palliative radiotherapy is allowed.

    For locally recurrent disease, the following treatment is allowed
    * Prior radiotherapy with curative intent
    * Prior chemo-radiotherapy with curative intent
    * Adjuvant chemotherapy
    * Localised palliative radiotherapy Prior chemotherapy must be > 6 months before screening
12. Severe intercurrent infections
13. Prior immunotherapy for metastatic or locally recurrent disease

The following is allowable:

• Adjuvant immunotherapy/ biologics Prior adjuvant immunotherapy/ biologics must be > 6 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Chong TOH, Study Chair — National Cancer Centre Singapore (NCCS)
Locations (30):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California Davis Health, Sacramento, California
  - UCSF HDF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baylor Scott & White, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Malaysia (7):
  - Site MY-03, George Town, Pulau Pinang
  - Site MY-06, George Town, Pulau Pinang
  - Site MY-07, Johor Bahru
  - Site MY-01, Kuala Lumpur
  - Site MY-04, Kuala Lumpur
  - Site MY-05, Kuala Lumpur
  - Site MY-08, Kuala Lumpur
- Singapore (2):
  - Site SG-11, Singapore
  - Site SG-12, Singapore
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (7):
  - Site TH-42, Bangkok
  - Site TH-43, Bangkok
  - Site TH-41, Chiang Mai
  - Site TH-44, Khon Kaen
  - Site TH-47, Lopburi
  - Site TH-45, Ubon Ratchathani
  - Site TH-46, Udon Thani

REFERENCES:
- [Derived] Toh HC, Yang MH, Wang HM, Hsieh CY, Chitapanarux I, Ho KF, Hong RL, Ang MK, Colevas AD, Sirachainan E, Lertbutsayanukul C, Ho GF, Nadler E, Algazi A, Lulla P, Wirth LJ, Wirasorn K, Liu YC, Ang SF, Low SHJ, Tho LM, Hasbullah HH, Brenner MK, Wang WW, Ong WS, Tan SH, Horak I, Ding C, Myo A, Samol J. Gemcitabine, carboplatin, and Epstein-Barr virus-specific autologous cytotoxic T lymphocytes for recurrent or metastatic nasopharyngeal carcinoma: VANCE, an international randomized phase III trial. Ann Oncol. 2024 Dec;35(12):1181-1190. doi: 10.1016/j.annonc.2024.08.2344. Epub 2024 Sep 4. PMID 39241963
- See also: Sponsor — http://www.tessatherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized 330 subjects at 23 sites in Asia and 7 sites in the United States from 17 Jul 2014 to 28 Feb 2022.
Pre-assignment Details: Subjects were randomized in a 1:1 ratio to receive open-label Gemcitabine and Carpoblatin followed by Autologus Epstein-Barr Virus-specific Cytotoxic T Cells (Chemo + EBV-CTL) versus Gemcitabine and Carboplatin alone (Chemo Only).
Groups:
- Chemo + EBV-CTL: Two consecutive stages:
  * 4 cycles of combination IV gemcitabine (1000 mg/m2) and IV carboplatin (AUC2) on Days 1, 8, 15 every 28 days. Option to add 1 to 2 cycles (i.e., up to 6 cycles total)
  * 6 cycles of immunotherapy with EBV-specific CTL (1 x 10^8 cells/m2) starting 2 to 4 weeks after last chemotherapy treatment. Subsequent chemotherapy cycles occurred 2 weeks after the first immunotherapy dose, 6 weeks after the second immunotherapy dose, and every 8 weeks thereafter
- Chemo Only: 6 cycles of combination IV gemcitabine (1000 mg/m2) and IV carboplatin (AUC2) on Days 1, 8, 15 every 28 days.
Period: Overall Study
Arm/Group | Chemo + EBV-CTL | Chemo Only
Started | 164 | 166
Treatment Received: Gemcitabine/ Carboplatin | 163 | 162
Treatment Received: EBV-CTL | 133 | 0
Completed | 55 | 99
Not Completed | 109 | 67
Not completed — Adverse Event | 5 | 15
Not completed — Death | 16 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 14 | 7
Not completed — Progressive Disease | 69 | 21
Not completed — No Study Drug | 2 | 0
Not completed — Randomized by Mistake with Study Treatment | 0 | 1
Not completed — Non-compliance with Study Schedule | 1 | 0
Not completed — Other | 1 | 10
Not completed — Not treated | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Analysis Set - all subjects randomized to treatment.
Groups:
- Chemo + EBV-CTL: gemcitabine/carboplatin and EBV-CTL
- Chemo Only: gemcitabine/carboplatin
- Total: Total of all reporting groups
Arm/Group | Chemo + EBV-CTL | Chemo Only | Total
Number analyzed (Participants) | 164 | 166 | 330
Age, Continuous [Median (Full Range); unit: years] | 53 [30 to 80] | 55 [21 to 79] | 54 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 122 | 126 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 156 | 157 | 313
  Unknown or Not Reported | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 160 | 160 | 320
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 17 | 17 | 34
  United States | 14 | 15 | 29
  Taiwan | 34 | 34 | 68
  Malaysia | 53 | 53 | 106
  Thailand | 46 | 47 | 93
Nasopharyngeal Cancer (NPC) stage at time of study entry [Count of Participants; unit: Participants] — NPC staging by Investigator per 7th American Joint Committee on Cancer (AJCC); Tumor (T)1 Nasopharynx, oropharynx, nasal cavity without extension, T2 Parapharyngeal extension, T3 Skull base, paranasal sinuses, T4 Intracranial, cranial, hypopharynx, orbit, infratemporal fossa/masticator; Nodes (N)0 No lymph node metastasis, N1 Cervical, retropharyngeal nodes, ≤6 cm, N2 Bilateral metastasis, ≤6cm, N3 >6 cm, supraclavicular fossa, Metastasis (M)0 No metastasis, M1 metastasis. Stage II:T2 N0-1 M0, T1 N1 M0; Stage III:T1-3 N2 M0, T3 N0-1 M0; Stage IVA:T4 N0-2 M0; Stage IVB:T N3 M0; Stage IVC:T N M1
  Participants
    Stage II | 15 | 5 | 20
    Stage III | 15 | 16 | 31
    Stage IVA | 14 | 24 | 38
    Stage IVB | 23 | 34 | 57
    Stage IVC | 94 | 84 | 178
    Others | 3 | 3 | 6
Disease Status per Randomization Stratification [Count of Participants; unit: Participants]
  Metastatic | 115 | 116 | 231
  Locally recurrent | 49 | 50 | 99
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS Scale, as assessed by Investigator - Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG PS 0 | 87 | 99 | 186
    ECOG PS 1 | 73 | 65 | 138
    ECOG PS 2 | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Subjects With Advanced Nasopharyngeal Carcinoma.
Description: Efficacy of EBV-CTL following first line chemotherapy was compared to chemotherapy alone in terms of OS of subjects with advanced nasopharyngeal carcinoma. Overall survival was defined as the duration in months from the day of randomization until death from any cause for a subject known to be deceased, or censored at the last contact date that a subject was known to be alive or lost to follow-up.
Time Frame: From randomization until death, assessed up to 7 years. Survivors and lost to follow-up subjects were censored at the date of last contact. Survival follow-up was done every 12 weeks from end of treatment.
Population: Intent-to-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Chemo + EBV-CTL: gemcitabine+carboplatin and EBV-CTL
- Chemo Only: gemcitabine+carboplatin
Arm/Group | Chemo + EBV-CTL | Chemo Only
Number analyzed (Participants) | 164 | 166
Months | 25 [19.7 to 31.8] | 24.9 [19.7 to 32.8]
Statistical Analysis 1: Comparison: Chemo + EBV-CTL vs Chemo Only; Test type: Superiority; p = 0.1942, Log Rank — Between-treatment comparisons were assessed using stratified log-rank test stratified by country and disease stage per randomization stratification; Log-rank test of Hazards Ration equals 1, using Cox proportional hazards regression; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.91 to 1.56] — Hazard ratios were estimated using Cox proportional hazards regression

2. Secondary Outcome: Progression-free Survival (PFS) of Subjects With Advanced Nasopharyngeal Carcinoma.
Description: Progression-free survival was defined as the duration from randomization to the first occurrence of documented disease progression [based on imaging results] or death from any cause, whichever occurred first.
Time Frame: From randomization until first occurrence of disease progression or death of any cause, whichever occurred first, assessed up to 7 years. Subjects who received subsequent anti-cancer therapy were censored at the date of last tumor assessment.
Population: Intent-to-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemo + EBV-CTL | Chemo Only
Number analyzed (Participants) | 164 | 166
Months | 7.9 [7.1 to 8.2] | 8.5 [8.1 to 9.6]

3. Secondary Outcome: Overall Response Rate (ORR) of Subjects With Advanced Nasopharyngeal Carcinoma.
Description: Overall response rate was assessed by sites using computed tomography/magnetic resonance imaging based on RECIST version 1.1, which defined Complete Response (CR) as disappearance of all lesions and pathologic lymph nodes; Partial Response (PR) as >=30% decrease in the sum of the longest diameter (SLD) of target lesions, no new lesions, no progression of non-target lesions; Stable disease (SD) as no PR and no progressive disease (PD); PD as >=20% increase SLD compared to smallest SLD or progression of non-target lesions or new lesions. The ORR for each treatment arm was comprised of the proportion of subjects who achieved a best overall response of CR or PR while on treatment (until End of Treatment visit), taking as reference the tumor measurement at baseline. Subjects who achieved CR or PR are responders, otherwise are non-responders.
Time Frame: From randomization until End of Treatment, an average of 13 months for the gemcitabine+carboplatin and EBVCTL arm and 6 months for the gemcitabine+carboplatin only arm.
Population: Intent-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo + EBV-CTL | Chemo Only
Number analyzed (Participants) | 164 | 166
Participants
  Responders (CR/PR) | 100 | 105
  Non-Responders (SD/PD/NA/NE) | 64 | 61

4. Secondary Outcome: Clinical Benefit Rate (CBR) of Subjects With Advanced Nasopharyngeal Carcinoma.
Description: Clinical benefit rate (CBR) was assessed using computed tomography/magnetic resonance imaging based on RECIST version 1.1., which defined CR as disappearance of all lesions and pathologic lymph nodes; PR as >=30% decrease in the sum of the longest diameter (SLD) of target lesions, no new lesions, no progression of non-target lesions; SD as no PR and no PD; PD as >=20% increase SLD compared to smallest SLD or progression of non-target lesions or new lesions. CBR was defined as the proportion of subjects who achieved CR, PR, or SD while on treatment (until End of Treatment visit), taking as reference the tumor measurement at baseline.
Time Frame: as for outcome 3
Population: Intent-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo + EBV-CTL | Chemo Only
Number analyzed (Participants) | 164 | 166
Participants
  Clinical Benefit (CR/PR/2 consecutive SD) | 139 | 136
  No Clinical Benefit (Otherwise) | 25 | 30

5. Secondary Outcome: Best Overall Response (BOR) of Subjects With Advanced Nasopharyngeal Carcinoma.
Description: Best overall response (BOR) was assessed using computed tomography/magnetic resonance imaging based on RECIST version 1.1., which defined CR as disappearance of all lesions and pathologic lymph nodes; PR as >=30% decrease in the sum of the longest diameter (SLD) of target lesions, no new lesions, no progression of non-target lesions; SD as no PR and no PD; PD as >=20% increase SLD compared to smallest SLD or progression of non-target lesions or new lesions. The BOR of each treatment arm consisted of CR, PR, SD, PD, NE, and NA while on treatment (until End of Treatment visit), taking as reference the tumor measurement at baseline. The ORR was comprised of the proportion of subjects who achieved a BOR of CR or PR.
Time Frame: as for outcome 3
Population: Intent-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo + EBV-CTL | Chemo Only
Number analyzed (Participants) | 164 | 166
Participants
  Complete Response (CR) | 6 | 14
  Partial Response (PR) | 94 | 91
  Stable Disease (SD) | 45 | 41
  Progressive Disease (PD) | 9 | 10
  NE (Not evaluable) | 1 | 0
  NA (Not applicable) | 9 | 10

ADVERSE EVENTS:
Time Frame: Adverse events during the entire trial duration were monitored/assessed from randomization to end of treatment (approximately 13 months for Chemo+EBV-CTL and 6 months for Chemo Only).
Description: Safety analyses are based on the Safety Analysis Set, defined as all randomized subjects who received at least one dose of study treatment. Subjects were analyzed according to the treatment actually received.
Groups:
- Chemo + EBV-CTL: gemcitabine+carboplatin + EBV-CTL
Arm/Group | Chemo + EBV-CTL | Chemo Only
All-Cause Mortality (participants affected / at risk) | 16/163 | 8/162
Serious Adverse Events (participants affected / at risk) | 68/163 | 46/162
Other Adverse Events (participants affected / at risk) | 163/163 | 162/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo + EBV-CTL (N=163) | Chemo Only (N=162)
Pneumonia (Infections and infestations) | 9 | 8
Anemia (Blood and lymphatic system disorders) | 9 | 6
febrile neutropenia (Blood and lymphatic system disorders) | 5 | 4
Pyrexia (General disorders) | 7 | 4
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 6
Hyponatremia (Metabolism and nutrition disorders) | 10 | 2
Septic shock (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 1 | 2
Injection site infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 3
Bacteremia (Infections and infestations) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Blood disorder (Blood and lymphatic system disorders) | 1 | 0
Disease progression (General disorders) | 2 | 1
Death (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mouth hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Seizure (Nervous system disorders) | 3 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal hematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Platelet count decreased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Immune-mediated adverse reaction (Immune system disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo + EBV-CTL (N=163) | Chemo Only (N=162)
Anemia (Blood and lymphatic system disorders) | 111 | 101
Neutropenia (Blood and lymphatic system disorders) | 63 | 65
Thrombocytopenia (Blood and lymphatic system disorders) | 47 | 52
Leukopenia (Blood and lymphatic system disorders) | 39 | 49
Platelet count decreased (Investigations) | 61 | 81
Neutrophil count decreased (Investigations) | 59 | 66
White blood cell count decreased (Investigations) | 60 | 59
Alanine aminotransferase increased (Investigations) | 15 | 18
Aspartate aminotransferase increased (Investigations) | 16 | 13
Constipation (Gastrointestinal disorders) | 48 | 45
Nausea (Gastrointestinal disorders) | 24 | 31
Diarrhoea (Gastrointestinal disorders) | 18 | 21
Vomitting (Gastrointestinal disorders) | 16 | 13
Fatigue (General disorders) | 36 | 38
Pyrexia (General disorders) | 43 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Headache (Nervous system disorders) | 23 | 18
Dizziness (Nervous system disorders) | 18 | 15
Hypoaesthesia (Nervous system disorders) | 9 | 8
Pneumonia (Infections and infestations) | 10 | 10
Pruritis (Skin and subcutaneous tissue disorders) | 14 | 21
Rash (Skin and subcutaneous tissue disorders) | 16 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 23 | 15
Decreased appetite (Metabolism and nutrition disorders) | 19 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 11
Insomnia (Psychiatric disorders) | 15 | 23
Tinnitus (Ear and labyrinth disorders) | 8 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT02578641/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT02578641/SAP_001.pdf